CLINICAL TRIAL: NCT00005680
Title: Whitehall II - Social and Occupational Influences On Health and Illness
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1070; R01HL036310 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Ischemia; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Ischemia; Hypertension

SUMMARY:
To examine the effect on health and disease of the work environment, psychological workload, control over work pacing and content, opportunity for use of skills, social support at work; the moderating effect on these relationships of social supports; and, the interaction between these psychosocial factors and other established risk factors in the etiology of chronic disease.

DETAILED DESCRIPTION:
BACKGROUND:

One of the major health problems facing industrialized countries is the persisting social class differences in the rate of occurrence of the major chronic diseases. It is true in the United States as it is in the United Kingdom, Scandinavia, Japan, and other countries. The advantage of investigating these social differences in the United Kingdom is that they have been most extensively documented, but findings are likely to be generalizable. The Black Report comprehensively reviewed the persisting social inequalities in health and concluded that the reasons were not completely understood. The Whitehall Study of the British civil service confirms the social gradient in mortality.

In the British civil service studies, as in the country as a whole, social class is defined on the basis of occupation. This raises the question as to whether the observed differences in morbidity and mortality are due to factors related to occupation or the general way of life. In many countries there are well documented social class differences in aspects of life-style: smoking, leisure-time physical activity, obesity, diet. Such differences were confirmed in civil servants studies, but these were insufficient to account for differences in mortality. There are thus two types of question: what accounts for the differences in smoking and other aspects of life style among men and women in different occupations? and; to what extent may the unexplained social differences in disease rates be related to factors associated with work as distinct from way of life?

DESIGN NARRATIVE:

There was a cross-sectional study and a short-term longitudinal study linking baseline data with morbidity based on sickness-absence records collected over an eighteen month period. Each subject was screened in an on-site work clinic. Questions were included on birthdate, civil service grade, marital status, family history of cardiovascular disease, occupation, car and house ownership, ethnicity, medical history of cardiovascular and respiratory problems, smoking, coffee and alcohol use, dietary intake, physical activity, work characteristics, social support, life satisfaction, life events, and mental illness. Type A behavior was assessed by the Framingham Type A Scale. A separately funded physical exam was conducted and included data on blood pressure, height, weight, pulse, ECG, blood clotting factors, and serum cholesterol. Initial analysis included calculation of prevalence rates of ischemic heart disease by age, sex, and social class as measured by employment grade. Dependent variables were crosstabulated for various categories of independent variables. The independent variables consisted of measures of psychosocial stress arising from work and personal situations.

The study was renewed in 1993 and again in 1997 to continue the follow-up of the cohort and collect further outcome data. This was achieved by 1) continued collection of sickness absence data; 2) obtaining information from GP's regarding long spells of absence; 3) obtaining death certificates and cancer registrations; and 4) a repeat questionnaire to all 10,314 participants to ensure completeness of outcome data. With additional outcome data the investigators used their extensive exposure database to explain the socio-economic gradient in health, encompassing both external influences and biomedical mechanisms. The main focus of the analysis was the role of work stress and social supports and networks both in explaining differences in health between socio-economic groups and individual differences in health. The analysis of these individual differences in health paid particular attention to women and ethnic minorities.

The study was renewed in 2002 to :(1) determine the extent to which socio-economic position and psychosocial factors influence pathophysiological responses and sub-clinical vascular disease directly and via health related behaviors, (2) examine psychosocial explanations for socio-economic differences in coronary health in an occupational cohort moving out of work, (3) determine, in our aging population, the relationships between socio-economic position, coronary disease and health functioning and disability.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marmot — University of London

REFERENCES:
- [Background] Stansfeld S, Marmot M. Deriving a survey measure of social support: the reliability and validity of the Close Persons Questionnaire. Soc Sci Med. 1992 Oct;35(8):1027-35. doi: 10.1016/0277-9536(92)90242-i. PMID 1411697
- [Background] Stansfeld SA, Marmot MG. Social class and minor psychiatric disorder in British Civil Servants: a validated screening survey using the General Health Questionnaire. Psychol Med. 1992 Aug;22(3):739-49. doi: 10.1017/s0033291700038186. PMID 1410098
- [Background] Pilgrim JA, Stansfeld S, Marmot M. Low blood pressure, low mood? BMJ. 1992 Jan 11;304(6819):75-8. doi: 10.1136/bmj.304.6819.75. PMID 1737142
- [Background] Marmot MG, Smith GD, Stansfeld S, Patel C, North F, Head J, White I, Brunner E, Feeney A. Health inequalities among British civil servants: the Whitehall II study. Lancet. 1991 Jun 8;337(8754):1387-93. doi: 10.1016/0140-6736(91)93068-k. PMID 1674771
- [Background] Rael EG, Stansfeld SA, Shipley M, Head J, Feeney A, Marmot M. Sickness absence in the Whitehall II study, London: the role of social support and material problems. J Epidemiol Community Health. 1995 Oct;49(5):474-81. doi: 10.1136/jech.49.5.474. PMID 7499989
- [Background] Marmot M, Feeney A, Shipley M, North F, Syme SL. Sickness absence as a measure of health status and functioning: from the UK Whitehall II study. J Epidemiol Community Health. 1995 Apr;49(2):124-30. doi: 10.1136/jech.49.2.124. PMID 7798038
- [Background] Stansfeld S, Feeney A, Head J, Canner R, North F, Marmot M. Sickness absence for psychiatric illness: the Whitehall II Study. Soc Sci Med. 1995 Jan;40(2):189-97. doi: 10.1016/0277-9536(94)e0064-y. PMID 7899931
- [Background] Roberts R, Brunner E, White I, Marmot M. Gender differences in occupational mobility and structure of employment in the British Civil Service. Soc Sci Med. 1993 Dec;37(12):1415-25. doi: 10.1016/0277-9536(93)90175-4. PMID 8303325
- [Background] Brunner EJ, Marmot MG, White IR, O'Brien JR, Etherington MD, Slavin BM, Kearney EM, Smith GD. Gender and employment grade differences in blood cholesterol, apolipoproteins and haemostatic factors in the Whitehall II study. Atherosclerosis. 1993 Sep;102(2):195-207. doi: 10.1016/0021-9150(93)90162-n. PMID 8251006
- [Background] Stansfeld SA, Smith GD, Marmot M. Association between physical and psychological morbidity in the Whitehall II Study. J Psychosom Res. 1993 Apr;37(3):227-38. doi: 10.1016/0022-3999(93)90031-a. PMID 8478817
- [Background] Marmot MG, North F, Feeney A, Head J. Alcohol consumption and sickness absence: from the Whitehall II study. Addiction. 1993 Mar;88(3):369-82. doi: 10.1111/j.1360-0443.1993.tb00824.x. PMID 8461854
- [Background] North F, Syme SL, Feeney A, Head J, Shipley MJ, Marmot MG. Explaining socioeconomic differences in sickness absence: the Whitehall II Study. BMJ. 1993 Feb 6;306(6874):361-6. doi: 10.1136/bmj.306.6874.361. PMID 8461681
- [Background] Marmot M. Social determinants of health: from observation to policy. Med J Aust. 2000 Apr 17;172(8):379-82. doi: 10.5694/j.1326-5377.2000.tb124011.x. PMID 10840490
- [Background] Kumari M, Brunner E, Fuhrer R. Minireview: mechanisms by which the metabolic syndrome and diabetes impair memory. J Gerontol A Biol Sci Med Sci. 2000 May;55(5):B228-32. doi: 10.1093/gerona/55.5.b228. PMID 10819309
- [Background] Fuhrer R, Head J, Marmot MG. Social position, age, and memory performance in the Whitehall II Study. Ann N Y Acad Sci. 1999;896:359-62. doi: 10.1111/j.1749-6632.1999.tb08141.x. No abstract available. PMID 10681922
- [Background] Brunner E, Shipley MJ, Blane D, Smith GD, Marmot MG. When does cardiovascular risk start? Past and present socioeconomic circumstances and risk factors in adulthood. J Epidemiol Community Health. 1999 Dec;53(12):757-64. doi: 10.1136/jech.53.12.757. PMID 10656084
- [Background] Stansfeld S, Head J, Ferrie J. Short-term disability, sickness absence, and social gradients in the Whitehall II Study. Int J Law Psychiatry. 1999 Sep-Dec;22(5-6):425-39. doi: 10.1016/s0160-2527(99)00019-9. No abstract available. PMID 10637751
- [Background] Stansfeld SA, Fuhrer R, Shipley MJ, Marmot MG. Work characteristics predict psychiatric disorder: prospective results from the Whitehall II Study. Occup Environ Med. 1999 May;56(5):302-7. doi: 10.1136/oem.56.5.302. PMID 10472303
- [Background] Martikainen P, Stansfeld S, Hemingway H, Marmot M. Determinants of socioeconomic differences in change in physical and mental functioning. Soc Sci Med. 1999 Aug;49(4):499-507. doi: 10.1016/s0277-9536(99)00135-5. PMID 10414809
- [Background] Hemingway H, Shipley M, Stansfeld S, Shannon H, Frank J, Brunner E, Marmot M. Are risk factors for atherothrombotic disease associated with back pain sickness absence? The Whitehall II Study. J Epidemiol Community Health. 1999 Apr;53(4):197-203. doi: 10.1136/jech.53.4.197. PMID 10396544
- [Background] Hemingway H, Marmot M. Evidence based cardiology: psychosocial factors in the aetiology and prognosis of coronary heart disease. Systematic review of prospective cohort studies. BMJ. 1999 May 29;318(7196):1460-7. doi: 10.1136/bmj.318.7196.1460. No abstract available. PMID 10346775
- [Background] Nicholson A, White IR, Macfarlane P, Brunner E, Marmot M. Rose questionnaire angina in younger men and women: gender differences in the relationship to cardiovascular risk factors and other reported symptoms. J Clin Epidemiol. 1999 Apr;52(4):337-46. doi: 10.1016/s0895-4356(99)00007-4. PMID 10235174
- [Background] Martikainen PT, Marmot MG. Socioeconomic differences in weight gain and determinants and consequences of coronary risk factors. Am J Clin Nutr. 1999 Apr;69(4):719-26. doi: 10.1093/ajcn/69.4.719. PMID 10197574
- [Background] Fuhrer R, Stansfeld SA, Chemali J, Shipley MJ. Gender, social relations and mental health: prospective findings from an occupational cohort (Whitehall II study). Soc Sci Med. 1999 Jan;48(1):77-87. doi: 10.1016/s0277-9536(98)00290-1. PMID 10048839
- [Background] Whitty CJ, Brunner EJ, Shipley MJ, Hemingway H, Marmot MG. Differences in biological risk factors for cardiovascular disease between three ethnic groups in the Whitehall II study. Atherosclerosis. 1999 Feb;142(2):279-86. doi: 10.1016/s0021-9150(98)00239-1. PMID 10030378
- [Background] Bosma H, Stansfeld SA, Marmot MG. Job control, personal characteristics, and heart disease. J Occup Health Psychol. 1998 Oct;3(4):402-9. doi: 10.1037//1076-8998.3.4.402. PMID 9805284
- [Background] Stafford M, Hemingway H, Stansfeld SA, Brunner E, Marmot M. Behavioural and biological correlates of physical functioning in middle aged office workers: the UK whitehall II study. J Epidemiol Community Health. 1998 Jun;52(6):353-8. doi: 10.1136/jech.52.6.353. PMID 9764255
- [Background] Stansfeld SA, Fuhrer R, Shipley MJ. Types of social support as predictors of psychiatric morbidity in a cohort of British Civil Servants (Whitehall II Study). Psychol Med. 1998 Jul;28(4):881-92. doi: 10.1017/s0033291798006746. PMID 9723143
- [Background] Stansfeld SA, Bosma H, Hemingway H, Marmot MG. Psychosocial work characteristics and social support as predictors of SF-36 health functioning: the Whitehall II study. Psychosom Med. 1998 May-Jun;60(3):247-55. doi: 10.1097/00006842-199805000-00004. PMID 9625210
- [Background] Feeney A, North F, Head J, Canner R, Marmot M. Socioeconomic and sex differentials in reason for sickness absence from the Whitehall II Study. Occup Environ Med. 1998 Feb;55(2):91-8. doi: 10.1136/oem.55.2.91. PMID 9614392
- [Background] Bosma H, Peter R, Siegrist J, Marmot M. Two alternative job stress models and the risk of coronary heart disease. Am J Public Health. 1998 Jan;88(1):68-74. doi: 10.2105/ajph.88.1.68. PMID 9584036
- [Background] Stafford M, Hemingway H, Marmot M. Current obesity, steady weight change and weight fluctuation as predictors of physical functioning in middle aged office workers: the Whitehall II Study. Int J Obes Relat Metab Disord. 1998 Jan;22(1):23-31. doi: 10.1038/sj.ijo.0800539. PMID 9481596
- [Background] Stansfeld SA, Head J, Marmot MG. Explaining social class differences in depression and well-being. Soc Psychiatry Psychiatr Epidemiol. 1998 Jan;33(1):1-9. doi: 10.1007/s001270050014. PMID 9448438
- [Background] Stallone DD, Brunner EJ, Bingham SA, Marmot MG. Dietary assessment in Whitehall II: the influence of reporting bias on apparent socioeconomic variation in nutrient intakes. Eur J Clin Nutr. 1997 Dec;51(12):815-25. doi: 10.1038/sj.ejcn.1600491. PMID 9426356
- [Background] Hemingway H, Stafford M, Stansfeld S, Shipley M, Marmot M. Is the SF-36 a valid measure of change in population health? Results from the Whitehall II Study. BMJ. 1997 Nov 15;315(7118):1273-9. doi: 10.1136/bmj.315.7118.1273. PMID 9390054
- [Background] Brunner EJ, Marmot MG, Nanchahal K, Shipley MJ, Stansfeld SA, Juneja M, Alberti KG. Social inequality in coronary risk: central obesity and the metabolic syndrome. Evidence from the Whitehall II study. Diabetologia. 1997 Nov;40(11):1341-9. doi: 10.1007/s001250050830. PMID 9389428
- [Background] Armstrong NC, Paganga G, Brunner E, Miller NJ, Nanchahal K, Shipley M, Rice-Evans CA, Marmot MG, Diplock AT. Reference values for alpha-tocopherol and beta-carotene in the Whitehall II Study. Free Radic Res. 1997 Aug;27(2):207-19. doi: 10.3109/10715769709097853. PMID 9350425
- [Background] Sheffield D, Smith GD, Carroll D, Shipley MJ, Marmot MG. The effects of blood pressure resting level and lability on cardiovascular reactions to laboratory stress. Int J Psychophysiol. 1997 Sep;27(2):79-86. doi: 10.1016/s0167-8760(97)00044-5. PMID 9342639
- [Background] Hemingway H, Nicholson A, Stafford M, Roberts R, Marmot M. The impact of socioeconomic status on health functioning as assessed by the SF-36 questionnaire: the Whitehall II Study. Am J Public Health. 1997 Sep;87(9):1484-90. doi: 10.2105/ajph.87.9.1484. PMID 9314801
- [Background] Marmot MG, Bosma H, Hemingway H, Brunner E, Stansfeld S. Contribution of job control and other risk factors to social variations in coronary heart disease incidence. Lancet. 1997 Jul 26;350(9073):235-9. doi: 10.1016/s0140-6736(97)04244-x. PMID 9242799
- [Background] Stansfeld SA, Fuhrer R, Head J, Ferrie J, Shipley M. Work and psychiatric disorder in the Whitehall II Study. J Psychosom Res. 1997 Jul;43(1):73-81. doi: 10.1016/s0022-3999(97)00001-9. PMID 9263933
- [Background] Stansfeld SA, Roberts R, Foot SP. Assessing the validity of the SF-36 General Health Survey. Qual Life Res. 1997 Apr;6(3):217-24. doi: 10.1023/a:1026406620756. PMID 9226979
- [Background] Carroll D, Davey Smith G, Sheffield D, Shipley MJ, Marmot MG. The relationship between socioeconomic status, hostility, and blood pressure reactions to mental stress in men: data from the Whitehall II study. Health Psychol. 1997 Mar;16(2):131-6. doi: 10.1037//0278-6133.16.2.131. PMID 9269883
- [Background] Hemingway H, Shipley MJ, Stansfeld S, Marmot M. Sickness absence from back pain, psychosocial work characteristics and employment grade among office workers. Scand J Work Environ Health. 1997 Apr;23(2):121-9. doi: 10.5271/sjweh.189. PMID 9167235
- [Background] Marmot M, Ryff CD, Bumpass LL, Shipley M, Marks NF. Social inequalities in health: next questions and converging evidence. Soc Sci Med. 1997 Mar;44(6):901-10. doi: 10.1016/s0277-9536(96)00194-3. PMID 9080570
- [Background] Bosma H, Marmot MG, Hemingway H, Nicholson AC, Brunner E, Stansfeld SA. Low job control and risk of coronary heart disease in Whitehall II (prospective cohort) study. BMJ. 1997 Feb 22;314(7080):558-65. doi: 10.1136/bmj.314.7080.558. PMID 9055714
- [Background] Brunner E, Davey Smith G, Marmot M, Canner R, Beksinska M, O'Brien J. Childhood social circumstances and psychosocial and behavioural factors as determinants of plasma fibrinogen. Lancet. 1996 Apr 13;347(9007):1008-13. doi: 10.1016/s0140-6736(96)90147-6. PMID 8606563
- [Background] North FM, Syme SL, Feeney A, Shipley M, Marmot M. Psychosocial work environment and sickness absence among British civil servants: the Whitehall II study. Am J Public Health. 1996 Mar;86(3):332-40. doi: 10.2105/ajph.86.3.332. PMID 8604757
- [Background] Roberts R, Brunner E, Marmot M. Psychological factors in the relationship between alcohol and cardiovascular morbidity. Soc Sci Med. 1995 Dec;41(11):1513-6. doi: 10.1016/0277-9536(95)00056-d. PMID 8607042
- [Background] Carroll D, Smith GD, Sheffield D, Shipley MJ, Marmot MG. Pressor reactions to psychological stress and prediction of future blood pressure: data from the Whitehall II Study. BMJ. 1995 Mar 25;310(6982):771-6. doi: 10.1136/bmj.310.6982.771. PMID 7711581
- [Background] Marmot M, Shipley M, Brunner E, Hemingway H. Relative contribution of early life and adult socioeconomic factors to adult morbidity in the Whitehall II study. J Epidemiol Community Health. 2001 May;55(5):301-7. doi: 10.1136/jech.55.5.301. PMID 11297647
- [Background] Ferrie JE, Martikainen P, Shipley MJ, Marmot MG, Stansfeld SA, Smith GD. Employment status and health after privatisation in white collar civil servants: prospective cohort study. BMJ. 2001 Mar 17;322(7287):647-51. doi: 10.1136/bmj.322.7287.647. PMID 11250849
- [Background] Ferrie JE, Shipley MJ, Marmot MG, Martikainen P, Stansfeld SA, Smith GD. Job insecurity in white-collar workers: toward an explanation of associations with health. J Occup Health Psychol. 2001 Jan;6(1):26-42. doi: 10.1037//1076-8998.6.1.26. PMID 11199254
- [Background] Mein G, Martikainen P, Stansfeld SA, Brunner EJ, Fuhrer R, Marmot MG. Predictors of early retirement in British civil servants. Age Ageing. 2000 Nov;29(6):529-36. doi: 10.1093/ageing/29.6.529. PMID 11191246
- [Background] Kumari M, Marmot M, Brunner E. Social determinants of von willebrand factor: the Whitehall II study. Arterioscler Thromb Vasc Biol. 2000 Jul;20(7):1842-7. doi: 10.1161/01.atv.20.7.1842. PMID 10894827
- [Background] Carroll D, Smith GD, Shipley MJ, Steptoe A, Brunner EJ, Marmot MG. Blood pressure reactions to acute psychological stress and future blood pressure status: a 10-year follow-up of men in the Whitehall II study. Psychosom Med. 2001 Sep-Oct;63(5):737-43. doi: 10.1097/00006842-200109000-00006. PMID 11573021
- [Background] Hemingway H, Whitty CJ, Shipley M, Stansfeld MS, Brunner E, Fuhrer R, Marmot M. Psychosocial risk factors for coronary disease in White, South Asian and Afro-Caribbean civil servants: the Whitehall II study. Ethn Dis. 2001 Autumn;11(3):391-400. PMID 11572405
- [Background] Brunner E, Stallone D, Juneja M, Bingham S, Marmot M. Dietary assessment in Whitehall II: comparison of 7 d diet diary and food-frequency questionnaire and validity against biomarkers. Br J Nutr. 2001 Sep;86(3):405-14. doi: 10.1079/bjn2001414. PMID 11570993
- [Background] Martikainen P, Ishizaki M, Marmot MG, Nakagawa H, Kagamimori S. Socioeconomic differences in behavioural and biological risk factors: a comparison of a Japanese and an English cohort of employed men. Int J Epidemiol. 2001 Aug;30(4):833-8. doi: 10.1093/ije/30.4.833. PMID 11511613
- [Background] Stafford M, Bartley M, Mitchell R, Marmot M. Characteristics of individuals and characteristics of areas: investigating their influence on health in the Whitehall II study. Health Place. 2001 Jun;7(2):117-29. doi: 10.1016/s1353-8292(01)00004-1. PMID 11470225
- [Background] Brunner EJ, Wunsch H, Marmot MG. What is an optimal diet? Relationship of macronutrient intake to obesity, glucose tolerance, lipoprotein cholesterol levels and the metabolic syndrome in the Whitehall II study. Int J Obes Relat Metab Disord. 2001 Jan;25(1):45-53. doi: 10.1038/sj.ijo.0801543. PMID 11244457
- [Background] Ferrie JE, Shipley MJ, Stansfeld SA, Marmot MG. Effects of chronic job insecurity and change in job security on self reported health, minor psychiatric morbidity, physiological measures, and health related behaviours in British civil servants: the Whitehall II study. J Epidemiol Community Health. 2002 Jun;56(6):450-4. doi: 10.1136/jech.56.6.450. PMID 12011203
- [Background] Fuhrer R, Stansfeld SA. How gender affects patterns of social relations and their impact on health: a comparison of one or multiple sources of support from "close persons". Soc Sci Med. 2002 Mar;54(5):811-25. doi: 10.1016/s0277-9536(01)00111-3. PMID 11999495
- [Background] Griffin JM, Fuhrer R, Stansfeld SA, Marmot M. The importance of low control at work and home on depression and anxiety: do these effects vary by gender and social class? Soc Sci Med. 2002 Mar;54(5):783-98. doi: 10.1016/s0277-9536(01)00109-5. PMID 11999493
- [Background] Stansfeld SA, Fuhrer R, Shipley MJ, Marmot MG. Psychological distress as a risk factor for coronary heart disease in the Whitehall II Study. Int J Epidemiol. 2002 Feb;31(1):248-55. doi: 10.1093/ije/31.1.248. PMID 11914328
- [Background] Kuper H, Marmot M. Intimations of mortality: perceived age of leaving middle age as a predictor of future health outcomes within the Whitehall II study. Age Ageing. 2003 Mar;32(2):178-84. doi: 10.1093/ageing/32.2.178. PMID 12615561
- [Background] Singh-Manoux A, Clarke P, Marmot M. Multiple measures of socio-economic position and psychosocial health: proximal and distal measures. Int J Epidemiol. 2002 Dec;31(6):1192-9; discussion 1199-200. doi: 10.1093/ije/31.6.1192. PMID 12540721
- [Background] Kuper H, Marmot M. Job strain, job demands, decision latitude, and risk of coronary heart disease within the Whitehall II study. J Epidemiol Community Health. 2003 Feb;57(2):147-53. doi: 10.1136/jech.57.2.147. PMID 12540692
- [Background] Mein G, Martikainen P, Hemingway H, Stansfeld S, Marmot M. Is retirement good or bad for mental and physical health functioning? Whitehall II longitudinal study of civil servants. J Epidemiol Community Health. 2003 Jan;57(1):46-9. doi: 10.1136/jech.57.1.46. PMID 12490648
- [Background] Ferrie JE, Shipley MJ, Davey Smith G, Stansfeld SA, Marmot MG. Change in health inequalities among British civil servants: the Whitehall II study. J Epidemiol Community Health. 2002 Dec;56(12):922-6. doi: 10.1136/jech.56.12.922. PMID 12461113
- [Background] Brunner EJ, Hemingway H, Walker BR, Page M, Clarke P, Juneja M, Shipley MJ, Kumari M, Andrew R, Seckl JR, Papadopoulos A, Checkley S, Rumley A, Lowe GD, Stansfeld SA, Marmot MG. Adrenocortical, autonomic, and inflammatory causes of the metabolic syndrome: nested case-control study. Circulation. 2002 Nov 19;106(21):2659-65. doi: 10.1161/01.cir.0000038364.26310.bd. PMID 12438290
- [Background] Martikainen P, Brunner E, Marmot M. Socioeconomic differences in dietary patterns among middle-aged men and women. Soc Sci Med. 2003 Apr;56(7):1397-410. doi: 10.1016/s0277-9536(02)00137-5. PMID 12614692
- [Background] Stansfeld SA, Head J, Fuhrer R, Wardle J, Cattell V. Social inequalities in depressive symptoms and physical functioning in the Whitehall II study: exploring a common cause explanation. J Epidemiol Community Health. 2003 May;57(5):361-7. doi: 10.1136/jech.57.5.361. PMID 12700221
- [Background] Singh-Manoux A, Adler NE, Marmot MG. Subjective social status: its determinants and its association with measures of ill-health in the Whitehall II study. Soc Sci Med. 2003 Mar;56(6):1321-33. doi: 10.1016/s0277-9536(02)00131-4. PMID 12600368
- [Background] Ferrie JE, Shipley MJ, Stansfeld SA, Smith GD, Marmot M; Whitehall II Study. Future uncertainty and socioeconomic inequalities in health: the Whitehall II study. Soc Sci Med. 2003 Aug;57(4):637-46. doi: 10.1016/s0277-9536(02)00406-9. PMID 12821012
- [Background] Chandola T, Bartley M, Sacker A, Jenkinson C, Marmot M. Health selection in the Whitehall II study, UK. Soc Sci Med. 2003 May;56(10):2059-72. doi: 10.1016/s0277-9536(02)00201-0. PMID 12697197
- [Background] Hemingway H, Shipley M, Mullen MJ, Kumari M, Brunner E, Taylor M, Donald AE, Deanfield JE, Marmot M. Social and psychosocial influences on inflammatory markers and vascular function in civil servants (the Whitehall II study). Am J Cardiol. 2003 Oct 15;92(8):984-7. doi: 10.1016/s0002-9149(03)00985-8. PMID 14556880
- [Background] Rennie KL, Hemingway H, Kumari M, Brunner E, Malik M, Marmot M. Effects of moderate and vigorous physical activity on heart rate variability in a British study of civil servants. Am J Epidemiol. 2003 Jul 15;158(2):135-43. doi: 10.1093/aje/kwg120. PMID 12851226
- [Background] Head J, Stansfeld SA, Siegrist J. The psychosocial work environment and alcohol dependence: a prospective study. Occup Environ Med. 2004 Mar;61(3):219-24. doi: 10.1136/oem.2002.005256. PMID 14985516
- [Background] Chandola T, Kuper H, Singh-Manoux A, Bartley M, Marmot M. The effect of control at home on CHD events in the Whitehall II study: Gender differences in psychosocial domestic pathways to social inequalities in CHD. Soc Sci Med. 2004 Apr;58(8):1501-9. doi: 10.1016/S0277-9536(03)00352-6. PMID 14759693
- [Background] Siegrist J, Starke D, Chandola T, Godin I, Marmot M, Niedhammer I, Peter R. The measurement of effort-reward imbalance at work: European comparisons. Soc Sci Med. 2004 Apr;58(8):1483-99. doi: 10.1016/S0277-9536(03)00351-4. PMID 14759692
- [Background] Britton A, Marmot M. Different measures of alcohol consumption and risk of coronary heart disease and all-cause mortality: 11-year follow-up of the Whitehall II Cohort Study. Addiction. 2004 Jan;99(1):109-16. doi: 10.1111/j.1360-0443.2004.00530.x. PMID 14678069
- [Background] Dykes J, Brunner EJ, Martikainen PT, Wardle J. Socioeconomic gradient in body size and obesity among women: the role of dietary restraint, disinhibition and hunger in the Whitehall II study. Int J Obes Relat Metab Disord. 2004 Feb;28(2):262-8. doi: 10.1038/sj.ijo.0802523. PMID 14647173
- [Background] Singh-Manoux A, Richards M, Marmot M. Leisure activities and cognitive function in middle age: evidence from the Whitehall II study. J Epidemiol Community Health. 2003 Nov;57(11):907-13. doi: 10.1136/jech.57.11.907. PMID 14600119
- [Background] Singh-Manoux A, Britton AR, Marmot M. Vascular disease and cognitive function: evidence from the Whitehall II Study. J Am Geriatr Soc. 2003 Oct;51(10):1445-50. doi: 10.1046/j.1532-5415.2003.51464.x. PMID 14511166
- [Background] Kivimaki M, Head J, Ferrie JE, Shipley MJ, Vahtera J, Marmot MG. Sickness absence as a global measure of health: evidence from mortality in the Whitehall II prospective cohort study. BMJ. 2003 Aug 16;327(7411):364. doi: 10.1136/bmj.327.7411.364. PMID 12919985
- [Background] Rennie KL, McCarthy N, Yazdgerdi S, Marmot M, Brunner E. Association of the metabolic syndrome with both vigorous and moderate physical activity. Int J Epidemiol. 2003 Aug;32(4):600-6. doi: 10.1093/ije/dyg179. PMID 12913036
- [Background] Ferrie JE, Kivimaki M, Head J, Shipley MJ, Vahtera J, Marmot MG. A comparison of self-reported sickness absence with absences recorded in employers' registers: evidence from the Whitehall II study. Occup Environ Med. 2005 Feb;62(2):74-9. doi: 10.1136/oem.2004.013896. PMID 15657187
- [Background] Ferrie JE, Shipley MJ, Newman K, Stansfeld SA, Marmot M. Self-reported job insecurity and health in the Whitehall II study: potential explanations of the relationship. Soc Sci Med. 2005 Apr;60(7):1593-602. doi: 10.1016/j.socscimed.2004.08.006. PMID 15652690
- [Background] Kivimaki M, Head J, Ferrie JE, Hemingway H, Shipley MJ, Vahtera J, Marmot MG. Working while ill as a risk factor for serious coronary events: the Whitehall II study. Am J Public Health. 2005 Jan;95(1):98-102. doi: 10.2105/AJPH.2003.035873. PMID 15623867
- [Background] Marmot M, Brunner E. Cohort Profile: the Whitehall II study. Int J Epidemiol. 2005 Apr;34(2):251-6. doi: 10.1093/ije/dyh372. Epub 2004 Dec 2. No abstract available. PMID 15576467
- [Background] Talmud PJ, Lewis SJ, Hawe E, Martin S, Acharya J, Marmot MG, Humphries SE, Brunner EJ. No APOEepsilon4 effect on coronary heart disease risk in a cohort with low smoking prevalence: the Whitehall II study. Atherosclerosis. 2004 Nov;177(1):105-12. doi: 10.1016/j.atherosclerosis.2004.06.008. PMID 15488872
- [Background] Kivimaki M, Ferrie JE, Head J, Shipley MJ, Vahtera J, Marmot MG. Organisational justice and change in justice as predictors of employee health: the Whitehall II study. J Epidemiol Community Health. 2004 Nov;58(11):931-7. doi: 10.1136/jech.2003.019026. PMID 15483310
- [Background] Kumari M, Head J, Marmot M. Prospective study of social and other risk factors for incidence of type 2 diabetes in the Whitehall II study. Arch Intern Med. 2004 Sep 27;164(17):1873-80. doi: 10.1001/archinte.164.17.1873. PMID 15451762
- [Background] Bartley M, Martikainen P, Shipley M, Marmot M. Gender differences in the relationship of partner's social class to behavioural risk factors and social support in the Whitehall II study. Soc Sci Med. 2004 Nov;59(9):1925-36. doi: 10.1016/j.socscimed.2004.03.002. PMID 15312926
- [Background] Stafford M, Martikainen P, Lahelma E, Marmot M. Neighbourhoods and self rated health: a comparison of public sector employees in London and Helsinki. J Epidemiol Community Health. 2004 Sep;58(9):772-8. doi: 10.1136/jech.2003.015941. PMID 15310804
- [Background] Britton A, Singh-Manoux A, Marmot M. Alcohol consumption and cognitive function in the Whitehall II Study. Am J Epidemiol. 2004 Aug 1;160(3):240-7. doi: 10.1093/aje/kwh206. PMID 15257997
- [Background] Singh-Manoux A, Ferrie JE, Chandola T, Marmot M. Socioeconomic trajectories across the life course and health outcomes in midlife: evidence for the accumulation hypothesis? Int J Epidemiol. 2004 Oct;33(5):1072-9. doi: 10.1093/ije/dyh224. Epub 2004 Jul 15. PMID 15256527
- [Background] Britton A, Shipley M, Marmot M, Hemingway H. Does access to cardiac investigation and treatment contribute to social and ethnic differences in coronary heart disease? Whitehall II prospective cohort study. BMJ. 2004 Aug 7;329(7461):318. doi: 10.1136/bmj.38156.690150.AE. Epub 2004 Jul 5. PMID 15237088
- [Background] Steptoe A, Willemsen G. The influence of low job control on ambulatory blood pressure and perceived stress over the working day in men and women from the Whitehall II cohort. J Hypertens. 2004 May;22(5):915-20. doi: 10.1097/00004872-200405000-00012. PMID 15097230
- [Background] Kumari M, Seeman T, Marmot M. Biological predictors of change in functioning in the Whitehall II study. Ann Epidemiol. 2004 Apr;14(4):250-7. doi: 10.1016/j.annepidem.2003.09.011. PMID 15066604
- [Background] Kunz-Ebrecht SR, Kirschbaum C, Marmot M, Steptoe A. Differences in cortisol awakening response on work days and weekends in women and men from the Whitehall II cohort. Psychoneuroendocrinology. 2004 May;29(4):516-28. doi: 10.1016/s0306-4530(03)00072-6. PMID 14749096
- [Background] Ferrie JE, Martikainen P, Shipley MJ, Marmot MG. Self-reported economic difficulties and coronary events in men: evidence from the Whitehall II study. Int J Epidemiol. 2005 Jun;34(3):640-8. doi: 10.1093/ije/dyi063. Epub 2005 Apr 14. PMID 15831564
- [Background] Langenberg C, Shipley MJ, Batty GD, Marmot MG. Adult socioeconomic position and the association between height and coronary heart disease mortality: findings from 33 years of follow-up in the Whitehall Study. Am J Public Health. 2005 Apr;95(4):628-32. doi: 10.2105/2004.046219. PMID 15798120
- [Background] Hillsdon MM, Brunner EJ, Guralnik JM, Marmot MG. Prospective study of physical activity and physical function in early old age. Am J Prev Med. 2005 Apr;28(3):245-50. doi: 10.1016/j.amepre.2004.12.008. PMID 15766611
- [Background] Kumari M, Marmot M, Rumley A, Lowe G. Social, behavioral, and metabolic determinants of plasma viscosity in the Whitehall II Study. Ann Epidemiol. 2005 May;15(5):398-404. doi: 10.1016/j.annepidem.2005.01.004. PMID 15840554
- [Background] Singh-Manoux A, Ferrie JE, Lynch JW, Marmot M. The role of cognitive ability (intelligence) in explaining the association between socioeconomic position and health: evidence from the Whitehall II prospective cohort study. Am J Epidemiol. 2005 May 1;161(9):831-9. doi: 10.1093/aje/kwi109. PMID 15840615
- [Background] Chandola T, Siegrist J, Marmot M. Do changes in effort-reward imbalance at work contribute to an explanation of the social gradient in angina? Occup Environ Med. 2005 Apr;62(4):223-30. doi: 10.1136/oem.2004.016675. PMID 15778254
- [Background] Hemingway H, Shipley M, Brunner E, Britton A, Malik M, Marmot M. Does autonomic function link social position to coronary risk? The Whitehall II study. Circulation. 2005 Jun 14;111(23):3071-7. doi: 10.1161/CIRCULATIONAHA.104.497347. Epub 2005 Jun 6. PMID 15939818
- [Background] Mein GK, Shipley MJ, Hillsdon M, Ellison GT, Marmot MG. Work, retirement and physical activity: cross-sectional analyses from the Whitehall II study. Eur J Public Health. 2005 Jun;15(3):317-22. doi: 10.1093/eurpub/cki087. Epub 2005 Jun 7. PMID 15941745
- [Background] Kivimaki M, Ferrie JE, Brunner E, Head J, Shipley MJ, Vahtera J, Marmot MG. Justice at work and reduced risk of coronary heart disease among employees: the Whitehall II Study. Arch Intern Med. 2005 Oct 24;165(19):2245-51. doi: 10.1001/archinte.165.19.2245. PMID 16246990
- [Background] Eliassen AH, Colditz GA, Rosner B, Willett WC, Hankinson SE. Serum lipids, lipid-lowering drugs, and the risk of breast cancer. Arch Intern Med. 2005 Oct 24;165(19):2264-71. doi: 10.1001/archinte.165.19.2264. PMID 16246993
- [Background] Zhao JH, Brunner EJ, Kumari M, Singh-Manoux A, Hawe E, Talmud PJ, Marmot MG, Humphries SE. APOE polymorphism, socioeconomic status and cognitive function in mid-life--the Whitehall II longitudinal study. Soc Psychiatry Psychiatr Epidemiol. 2005 Jul;40(7):557-63. doi: 10.1007/s00127-005-0925-y. Epub 2005 Jul 15. PMID 16021346